CLINICAL TRIAL: NCT01445769
Title: An Open-label Assessment of an Alternative Dosing Strategy of Ruxolitinib in Patients With Primary Myelofibrosis, Post-polycythemia Vera Myelofibrosis, and Post-essential Thrombocythemia Myelofibrosis
Brief Title: Alternative Dosing Strategy of Ruxolitinib in Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18424-261
Record Dates: First submitted 2011-09-23; First posted 2011-10-04 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis
Keywords: Myelofibrosis; Primary Myelofibrosis; PMF; Post-Polycythemia Vera Myelofibrosis; PPV-MF; Post-Essential Thrombocythemia Myelofibrosis; PET-MF; Open label; Ruxolitinib; 18424; Jak inhibitor
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib (Experimental): Participants initially received ruxolitinib 10 mg twice a day (bid) for 24 weeks. Dose increases of 5 mg bid were possible at Weeks 12 and 18 up to a maximum dose of 20 mg bid.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib was provided as 5 mg tablets. Dose increases were only permitted at wks 12 & 18 for lack of efficacy. Increases were restricted to patients who didn't meet criteria for a dose hold over the prior 6 wks, had a platelet count ≥ 100 x 10^9/L at wk 12 or ≥ 150 x 10^9/L at wk 18, and had a self-reported PGIC score of 3 (minimally improved) to 7 (very much worse) OR the subject's palpable spleen length below the costal margin was reduced by less than 40% relative to Baseline. Dose increases were elective and not required. Subjects were permitted a dose increase of 5 mg BID to 15 mg BID at wk 12 and to a maximum of 20 mg BID at wk 18. The protocol required dose decreases for thrombocytopenia (platelets <100 x 10^9/L) or protocol-defined anemia (decline in hemoglobin of at least 2 g/dL to a level < 8 g/dL, development of transfusion dependence, or a 50% increase in transfusion requirements for transfusion dependent subjects).
  Other Names: INCB018424; INC424

SUMMARY:
The purpose of this study was to evaluate the effect of an alternative dosing strategy of ruxolitinib in subjects with primary myelofibrosis (PMF), post-polycythemia vera-myelofibrosis (PPV-MF) and post essential thrombocythemia-myelofibrosis (PET-MF) in order to minimize the development of anemia and thrombocytopenia.

DETAILED DESCRIPTION:
This pilot study was designed to explore an alternative dosing approach with the purpose of reducing anemia and thrombocytopenia. Subjects began dosing at 10 mg bid and had the opportunity for dose increases based on assessments of efficacy and overall hematologic status in a defined prior dosing interval. Dose increases were restricted to those patients who did not meet criteria for or have a dose hold over the prior 6 weeks, had a platelet count ≥100 x 10^9/L at week 12 or ≥150 x 10^9/L at week 18, and had a self-reported Patient's Global Impression of Change (PGIC) score of 3 (minimally improved) to 7 (very much worse) OR the subject's palpable spleen length below the costal margin had been reduced by less than 40% at that visit relative to Baseline. Dose increases were elective and not required. Subjects were permitted a dose increase of 5 mg BID to 15 mg BID at Week 12 and to a maximum of 20 mg BID at Week 18. There were also protocol-required dose decreases for thrombocytopenia (platelets <100 x 10^9/L) or protocol-defined anemia (decline in hemoglobin of at least 2 g/dL to a level < 8 g/dL, development of transfusion dependence, or a 50% increase in transfusion requirements for transfusion dependent subjects).This approach assumed that beginning at a low dose for initial therapy might have a positive impact on the rate of the initial hemoglobin decline and the nadir by decreasing the level of JAK-mediated inhibition of hematopoiesis. Specific dose modifications were described to minimize excursions of hemoglobin levels into the Grade 3 or Grade 4 range.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (PPV-MF), or Post-Essential Thrombocythemia Myelofibrosis (PET-MF) as confirmed by bone marrow biopsy.
* Must score at least 2 points on the Dynamic International Prognostic Scoring System (DIPSS) scale for prognostic risk factors.
* Peripheral blast count < 5% at both Screening and Baseline hematology assessments.
* Must discontinue all drugs used to treat underlying myelofibrosis (MF) disease no later than Day -1 (the day prior to starting ruxolitinib).
* Must have hemoglobin value ≥ 6.5 g/dL and be willing to receive blood transfusions.
* Platelet count ≥ 100*10^9/L.
* Must have a palpable spleen.

Exclusion Criteria:

* Inadequate liver or bone marrow reserves, end stage renal disease on dialysis, clinically significant concurrent infections requiring therapy, or unstable cardiac function.
* Invasive malignancies over the previous 5 years (except treated early stage carcinomas of the skin, completely resected intraepithelial carcinoma of the cervix, and completely resected papillary thyroid and follicular thyroid cancers).
* Splenic irradiation within 6 months prior to receiving the first dose of study medication.
* Life expectancy less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William V Williams, MD, Study Director — Incyte Corporation
Locations (21):
- United States (21):
  - Highland, California
  - La Jolla, California
  - Los Angeles, California
  - Jacksonville, Florida
  - Orange City, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Southfield, Michigan
  - Morristown, New Jersey
  - Armonk, New York
  - Hickory, North Carolina
  - Canton, Ohio
  - Hazleton, Pennsylvania
  - Hershey, Pennsylvania
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - San Antonio, Texas

REFERENCES:
- [Derived] Talpaz M, Erickson-Viitanen S, Hou K, Hamburg S, Baer MR. Evaluation of an alternative ruxolitinib dosing regimen in patients with myelofibrosis: an open-label phase 2 study. J Hematol Oncol. 2018 Aug 7;11(1):101. doi: 10.1186/s13045-018-0642-0. PMID 30086777

RESULTS

PARTICIPANT FLOW:
Groups:
- Ruxolitinib: Participants initially received ruxolitinib 10 mg twice a day (bid). Dose increases of 5 mg bid were permitted at Weeks 12 and 18 for subjects who did not meet criteria for or have a dose hold over the prior 6 weeks, had a platelet count ≥100 x 10^9/L at week 12 or ≥150 x 10^9/L at week 18, and had a self-reported Patients' Global Impression of Change (PGIC) score of 3 (minimally improved) to 7 (very much worse) OR the subject's palpable spleen length had been reduced by less than 40% at that visit relative to Baseline. The maximum dose was 15 mg BID at Week 12 and 20 mg bid at Week 18. There were also protocol-required dose decreases for protocol-defined anemia and thrombocytopenia.
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 45
Completed | 37
Not Completed | 8
Not completed — Consent Withdrawn | 2
Not completed — Disease Progression | 1
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All enrolled participants. Note that this was a pilot study which was not sufficiently powered.
Groups:
- Ruxolitinib: Participants initially received ruxolitinib 10 mg twice a day (bid). Dose increases of 5 mg bid were permitted at Weeks 12 and 18 for subjects who did not meet criteria for or have a dose hold over the prior 6 weeks, had a platelet count ≥ 100 x 10^9/L at week 12 or ≥ 150 x 10^9/L at week 18, and had a self-reported PGIC score of 3 (minimally improved) to 7 (very much worse) OR the subject's palpable spleen length had been reduced by less than 40% at that visit relative to Baseline. The maximum dose was 15 mg BID at Week 12 and 20 mg bid at Week 18. There were also protocol-required dose decreases for protocol-defined anemia and thrombocytopenia.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change From Baseline in Spleen Volume at Week 24
Description: Spleen volume was measured using magnetic resonance imaging (MRI) or computed tomography (CT) scan. The MRIs were read in the central imaging laboratory. Spleen volume was obtained by outlining the circumference of the organ and determining the volume using the technique of least squares. MRI was the preferred method for obtaining spleen volume data. CT scans were performed if the participant was not a candidate for MRI. The CT scans were processed by the same central laboratory used for MRIs. The same method (MRI or CT) was used for all visits for a given participant unless a new contraindication to the use of MRI (eg, pacemaker insertion) occurred.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All enrolled participants. Note that 2 subjects did not have the Week 24 MRI; one subject dropped out for disease progression and two withdrew consent prior to the Week 24 MRI. Thus 40 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Ruxolitinib: Participants initially received ruxolitinib 10 mg twice a day (bid). Dose increases of 5 mg bid were permitted at Weeks 12 and 18 for subjects who did not meet criteria for or have a dose hold over the prior 6 weeks, had a platelet count ≥100 x 10^9/L at week 12 or ≥150 x 10^9/L at week 18, and had a self-reported PGIC score of 3 (minimally improved) to 7 (very much worse) OR the subject's palpable spleen length had been reduced by less than 40% at that visit relative to Baseline. The maximum dose was 15 mg BID at Week 12 and 20 mg bid at Week 18. There were also protocol-required dose decreases for protocol-defined anemia and thrombocytopenia. Only the subjects who had Week 24 spleen volume data are summarized.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 40
Percentage change | -14.9 (21.06)

2. Primary Outcome: Median Percent Change From Baseline in Spleen Volume at Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Median (Full Range); unit: : Percentage change
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 40
: Percentage change | -17.3 [-54.2 to 58.5]

3. Secondary Outcome: Mean Percentage Change From Baseline in the Total Symptom Score at Week 24
Description: Symptoms of myelofibrosis were assessed using a symptom diary, the modified Myelofibrosis Symptom Assessment Form (MFSAF v2.0). Participants were issued a hand-held device to record answers to queries regarding 7 symptoms of myelofibrosis each night from Baseline through Week 24. Symptoms assessed included night sweats, itching, abdominal discomfort, pain under ribs on left, feeling of fullness (early satiety), muscle/bone pain, and inactivity. The daily total symptom score (TSS) was the sum of the first 6 individual symptom scores (each on a scale of 0-10). Inactivity was not included in the total score. The Baseline TSS was the mean of daily total symptom scores from the last 7 consecutive days prior to the first study dose and ranged from 0 to 60. The Week 24 TSS was the mean of the daily total symptom scores from the last 28 consecutive days prior to the Week 24 visit and ranged from 0 to 60. A higher score indicates worse symptoms. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All enrolled participants. Note that 3 subjects did not have the Week 24 TSS; one subject dropped out for disease progression and two withdrew consent prior to the Week 24 TSS assessment. Thus 39 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Ruxolitinib: Participants initially received ruxolitinib 10 mg twice a day (bid). Dose increases of 5 mg bid were permitted at Weeks 12 and 18 for subjects who did not meet criteria for or have a dose hold over the prior 6 weeks, had a platelet count ≥100 x 10^9/L at week 12 or ≥150 x 10^9/L at week 18, and had a self-reported PGIC score of 3 (minimally improved) to 7 (very much worse) OR the subject's palpable spleen length had been reduced by less than 40% at that visit relative to Baseline. The maximum dose was 15 mg BID at Week 12 and 20 mg bid at Week 18. There were also protocol-required dose decreases for protocol-defined anemia and thrombocytopenia.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 39
Percentage change | -34.3 (69.05)

4. Secondary Outcome: Median Percent Change From Baseline in the Total Symptom Score at Week 24
Description: Symptoms of myelofibrosis were assessed using a symptom diary, the modified MFSAF v2.0. Participants were issued a hand-held device to record answers to queries regarding 7 symptoms of myelofibrosis each night from Baseline through Week 24. Symptoms assessed included night sweats, itching, abdominal discomfort, pain under ribs on left, feeling of fullness (early satiety), muscle/bone pain, and inactivity. The daily TSS was the sum of the first 6 individual symptom scores (each on a scale of 0-10). Inactivity was not included in the total score. The Baseline total symptom score was the mean of daily total symptom scores from the last 7 consecutive days prior to the first study dose and ranged from 0 to 60. The Week 24 total symptom score was the mean of the daily total symptom scores from the last 28 consecutive days prior to the Week 24 visit and ranged from 0 to 60. A higher score indicates worse symptoms. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 39
Percentage change | -45.6 [-100.0 to 261.9]

5. Secondary Outcome: Percentage of Participants With a ≥ 35% Reduction From Baseline in Spleen Volume at Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 45
Percentage of participants | 15.6 [6.5 to 29.5]

6. Secondary Outcome: Percentage of Participants With a ≥ 10% Reduction From Baseline in Spleen Volume at Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 45
Percentage of participants | 57.8 [42.2 to 72.3]

7. Secondary Outcome: Percentage of Participants With a ≥ 50% Improvement From Baseline in Total Symptom Score at Week 24
Description: Symptoms of myelofibrosis were assessed using a symptom diary, the modified MFSAF v2.0. Participants were issued a hand-held device to record answers to queries regarding 7 symptoms of myelofibrosis each night from Baseline through Week 24. Symptoms assessed included night sweats, itching, abdominal discomfort, pain under ribs on left, feeling of fullness (early satiety), muscle/bone pain, and inactivity. The daily total symptom score was the sum of the first 6 individual symptom scores (each on a scale of 0-10). Inactivity was not included in the total score. The Baseline total symptom score was the mean of daily total symptom scores from the last 7 consecutive days prior to the first study dose and ranged from 0 to 60. The Week 24 total symptom score was the mean of the daily total symptom scores from the last 28 consecutive days prior to the Week 24 visit and ranged from 0 to 60. A higher score indicates worse symptoms. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 45
Percentage of participants | 40.0 [25.7 to 55.7]

8. Secondary Outcome: Mean Percentage Change From Baseline in Palpable Spleen Length at Week 24
Description: Spleen length was assessed by manual palpation. The edge of the spleen was determined by palpation and measured in centimeters, using a soft ruler, from the costal margin to the point of greatest splenic protrusion.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All enrolled participants. Note that one subject had a non-palpable spleen at baseline, one subject did not have the Week 24 spleen palpation performed; one subject dropped out for disease progression and two withdrew consent prior to the Week 24 spleen palpation. Thus 40 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 40
Percentage change | -47.6 (42.05)

9. Secondary Outcome: Median Percent Change From Baseline in Palpable Spleen Length at Week 24
Description: as for outcome 8
Time Frame: Baseline to Week 24
Population: as for outcome 8
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 40
Percentage change | -39.8 [-100.0 to 26.7]

10. Secondary Outcome: Percentage of Participants With a ≥ 50% Improvement From Baseline in Their Transfusion Status or With New Transfusion Independence Status for Those Participants Who Were Transfusion Dependent at Baseline
Description: Transfusion dependence at Baseline is defined as subjects who received ≥ 2 units of red blood cell product(s) in the 12 consecutive weeks prior to the date of first dose.
  Transfusion independence On-Study is defined as subjects who received 0 units of red blood cell products over any 12-week period after starting dosing with ruxolitinib.
  Improvement in transfusion dependence On-Study is defined as a 50% or greater reduction in the frequency of red blood cell transfusions over any 12-week period after starting dosing with ruxolitinib.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All enrolled participants who were transfusion dependent at baseline (n=15).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 15
Percentage of participants | 20.0 [4.3 to 48.1]

11. Secondary Outcome: Percentage of Participants With Clinically Notable Anemia
Description: Clinically Notable Anemia was a pre-specified safety parameter examined at Weeks 12, 18 and 24 and defined as: 1) New onset Grade 3 or higher anemia in subjects who are transfusion independent at Baseline, 2) New onset transfusion dependence in subjects who are transfusion independent at Baseline, defined as receipt of ≥ 2 units in ≤ a 12-week interval, 3) 50% increase in transfusions compared to Baseline in subjects who are transfusion dependent at Baseline.
Time Frame: Baseline to Weeks 12, 18 and 24
Population: Safety population: All participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 45
Percentage of participants
  Week 12 | 33.3
  Week 18: number analyzed (Participants) | 44
  Week 18 | 27.3
  Week 24: number analyzed (Participants) | 43
  Week 24 | 27.9

12. Secondary Outcome: Mean Percentage Change in Abdominal Symptom Scores at Week 24.
Description: Symptoms of myelofibrosis were assessed using a symptom diary, the modified MFSAF v2.0. Participants were issued a hand-held device to record answers to queries regarding 7 symptoms of myelofibrosis each night from Baseline through Week 24. The abdominal symptom score was the sum of 3 individual symptom scores (abdominal discomfort, pain under ribs on left side, and feeling of fullness [early satiety]), each on a scale of 0 to 10. A higher score indicates worse symptoms. A negative change score indicates improvement. The Baseline abdominal symptom score was the mean of daily abdominal symptom scores from the last 7 consecutive days prior to the first study dose and ranged from 0 to 30. The Week 24 abdominal symptom score was the mean of the daily abdominal symptom scores from the last 28 consecutive days prior to the Week 24 visit and ranged from 0 to 30.
Time Frame: Week 24
Population: Intent-to-treat population: All enrolled participants. Note that three subjects did not have the Week 24 TSS; one subject dropped out for disease progression and two withdrew consent prior to the Week 24 TSS assessment. Thus 39 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 39
Percentage change | -33.2 (69.83)

13. Secondary Outcome: Median Percentage Change in Abdominal Symptom Scores at Week 24.
Description: Symptoms of myelofibrosis were assessed using a symptom diary, the modified MFSAF v2.0. Participants were issued a hand-held device to record answers to queries regarding 7 symptoms of myelofibrosis each night from Baseline through Week 24. The abdominal symptom score was the sum of 3 individual symptom scores (abdominal discomfort, pain under ribs on left side, and feeling of fullness [early satiety]).
Time Frame: Week 24
Population: as for outcome 12
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 39
Percentage change | -50.5 [-100.0 to 219.0]

14. Secondary Outcome: Number of Participants With Grade 3 or Grade 4 Adverse Events
Time Frame: Baseline to the end of the study
Population: Safety population: All participants who took at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 45
participants
  Anemia (Grade 3) | 9
  Thrombocytopenia (Grade 3) | 1
  Umbilical hernia (Grade 3) | 1
  Cholelithiasis (Grade 3) | 1
  Blood creatine phosphokinase increased (Grade 3) | 1
  Blood triglycerides increased (Grade 3) | 1
  Lipase increased (Grade 3) | 1
  Dehydration (Grade 3) | 1
  Hyperkalaemia (Grade 3) | 1
  Hypermagnesaemia (Grade 3) | 1
  Dizziness (Grade 3) | 1
  Myelodysplastic syndrome (Grade 4) | 1

15. Other Pre Specified Outcome: Dose Distribution at Week 24
Description: Average Daily Dose for the last 28 days on study.
Time Frame: Week 24
Population: Intent-to-treat population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 45
participants
  0-5 mg | 2
  > 5-10 mg | 14
  > 10-20 mg | 12
  > 20-30 mg | 12
  > 30-40 mg | 5

ADVERSE EVENTS:
Time Frame: From the first dose of study medication through the Follow-Up Visit.
Description: Safety population: All participants who took at least 1 dose of study drug.
Arm/Group | Ruxolitinib
Serious Adverse Events (participants affected / at risk) | 2/45
Other Adverse Events (participants affected / at risk) | 42/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=45)
Cholelithiasis (Hepatobiliary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=45)
Anemia (Blood and lymphatic system disorders) | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 10
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 3
Contusion (Injury, poisoning and procedural complications) | 5
Decreased appetite (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Night sweats (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3

LIMITATIONS AND CAVEATS:
This was a single arm pilot study. The patient population differed from Phase III studies of ruxolitinib in myelofibrosis and therefore comparisons to standard dosing cannot be made from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.